CLINICAL TRIAL: NCT01080443
Title: Open Label Balanced Randomized Two-treatment Two-period Two-sequence Single Dose Two-way Crossover Oral Bioequivalence Study of Mycophenolate Mofetil Capsules 250 mg in Normal Healthy Adult Human Subjects Under Fasting Conditions
Brief Title: Bioequivalence Study of Mycophenolate Mofetil 250 mg Capsule Under Fasting Condition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Panacea Biotec Ltd (Industry)
Responsible Party: Dr. Arani Chatterjee, Panacea Biotec Ltd.
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 328-07
Record Dates: First submitted 2010-03-02; First posted 2010-03-04 (Estimated); Last update posted 2010-03-12 (Estimated); Status verified 2010-03

CONDITIONS: Healthy Volunteers
Keywords: Bioequivalence study in healthy volunteers
MeSH Terms: interventions — Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cellcept® 250 mg Capsule (Active Comparator)
  Interventions: Drug: Mycophenolate Mofetil Capsule 250 mg
- Mycophenolate Mofetil Capsule 250 mg (Experimental)
  Interventions: Drug: Mycophenolate Mofetil Capsule 250 mg

INTERVENTIONS:
Drug: Mycophenolate Mofetil Capsule 250 mg — Subjects will be administered either Test Product or Reference Product with 240 mL of water according to randomization schedule
  Other Names: Mycophenolate Mofetil Capsule

SUMMARY:
The objective of the study is to compare the bioavailability and characterise the pharmacokinetic profile of Mycophenolate mofetil 250 mg capsules Panacea Biotech Ltd, India and Cellcept® 250 mg capsules Mycophenolate mofetil capsule, Roche Labs Inc. New Jersey, USA in normal, healthy, adult human subjects under fasting conditions, and to assess the bioequivalence.

DETAILED DESCRIPTION:
48 +8 (stand-by) normal healthy adult subjects will be enrolled in the study. Subjects will be administered either the Test or the Reference Product with 240 mL of water in each period as per the randomization schedule. Subjects will fast for at least 10 hours prior to dose administration and for at least 4 hours post dose. Standardized meals will be provided in each study period. Water will not be accessible to the subjects 1 hour Predose and 2 hours Post dose in each period. A total of 28 blood samples will be withdrawn for pharmacokinetic profiling. The concentration of mycophenolate mofetil and mycophenolic acid will be quantitated using validated LC-MS / MS method.ANOVA, two one-sided tests for bioequivalence, power and ratio analysis for un-transformed and ln-transformed pharmacokinetic parameters Cmax, AUC0-t AUC0-inf will be computed and reported for Mycophenolic acid. Bioequivalence of the test product with that of the reference product under fasting conditions will be concluded if the 90% confidence interval falls within the acceptance range of 80.00-125.00% for ln-transformed pharmacokinetic parameters Cmax, AUC0-t and AUC0-inf for Mycophenolic acid.

ELIGIBILITY:
Inclusion Criteria:

* Normal, healthy human volunteers between 18 and 60 years of age (both inclusive) living in and around Ahmedabad city of western part of India.
* Having a Body Mass Index (BMI) between 18.5 and 24.9 (both inclusive), calculated as weight in kg / height in m2.
* Not having any significant diseases or clinically significant abnormal findings during screening, medical history, physical examination, laboratory evaluations, 12 - lead ECG and X-ray chest (postero-anterior view) recordings.
* Able to comply with study procedures, in the opinion of the Principal Investigator.
* Able to give written consent for participation in the trial.
* In case of female subjects they must be (A) Surgically sterilized at least 6 months prior to study participation or (B) Those who are of child bearing potential must be using a suitable and effective double barrier contraceptive method or intra urine devices during the study.

Exclusion Criteria:

* Known hypersensitivity or idiosyncratic reaction to Mycophenolate Mofetil or any related drug.
* Any disease or condition which might compromise the haemopoietic, renal, hepatic, endocrine, pulmonary, central nervous, cardiovascular, immunological, dermatological, gastrointestinal or any other body system.
* Ingestion of a medicine at any time in 14 days before the start of the study. In any such case subject selection will be at the discretion of the Principal Investigator / Medical Expert.
* Any history or presence of asthma (including aspirin induced asthma) or nasal polyp or nonsteroidal anti-inflammatory drug (NSAID) induced urticaria.
* A recent history of alcoholism (<2 years) or of moderate (180 mL / day) alcohol use, or consumption of alcohol within 48 hour prior to receiving study medicine.
* Smokers, who smoke 10 or more cigarettes per day and / or unable to abstain from smoking during the study.
* The presence of clinically significant abnormal laboratory values during screening.
* Use of any recreational drugs or history of drug addiction or testing positive in pre study drug scan.
* History of psychiatric disorders.
* A history of difficulty in donating blood.
* Donation of blood (1 unit or 350 mL) within 90 days prior to receiving the first dose of study medicine.

Note: In case the blood loss is ≤ 200 mL, subject may be dosed 60 days after blood donation.

* A positive hepatitis screen including hepatitis B surface antigen and anti-hepatitis C virus (HCV) antibodies.
* A positive test result for anti-HIV antibody and / or syphilis.
* The receipt of an investigational product or participation in a drug research study within a period of 90 days prior to the first dose of study medicine. Elimination half-life of the study drug should be taken into consideration for inclusion of the subject in the study.

Note: If subject had participated in a study in which blood loss is ≤ 200 mL, subject can be dosed 60 days after the last sample of previous study.

* An unusual diet, for whatever reason (e.g. low-sodium), for four weeks prior to receiving the study medication and throughout the subject's participation in the study. In any such case subject selection will be at the discretion of the Principal Investigator / Medical Expert.
* Pregnant females or Nursing mothers
* Testing positive in urine pregnancy test.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2008-06; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
To compare the bioavailability of Mycophenolate mofetil 250 mg capsules Panacea Biotec Ltd, India and Cellcept® 250 mg capsules Mycophenolate mofetil capsule, Roche Labs Inc. New Jersey, USA, and to assess the bioequivalence. | up to 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Pankaj K Jha, Principal Investigator — Lambda Therapeutic Research Ltd.
Locations (1):
- Lambda Therapeutic Research Ltd., Ahmedabad, Gujarat, India